CLINICAL TRIAL: NCT02960113
Title: Is the Application of Scopolamine Patch With or Without Intra-operative Acupressure Point P6 Stimulation More Effective Than Intra-operative Acupressure Point P6 Stimulation Alone?
Brief Title: Scopolamine Patch and Acupressure Point P6 Stimulation for Reduction of Nausea and Vomiting During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shaul Cohen, M.D., Director of Obstetric Anesthesia, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro20160000234
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Nausea; Vomiting; Satisfaction
Keywords: cesarean section; acupressure point p6; scopolamine patch
MeSH Terms: conditions — Nausea; Vomiting; Personal Satisfaction | interventions — Butylscopolammonium Bromide; Scopolamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- scopolamine patch (Experimental): Scopolamine patch will be placed on the skin behind the right ear 1 hour before initiation of the regional anesthesia for the duration of surgery.
  Interventions: Drug: scopolamine patch
- acupressure point P6 (Experimental): Acupressure point P6 stimulation will be placed on the distal right forearm just above the crest of the wrist.
  Interventions: Device: acupressure point P6
- scopolamine patch + acupressure point P6 (Experimental): Will receive both scopolamine patch and acupressure point P6 stimulation, as described above.
  Interventions: Drug: scopolamine patch; Device: acupressure point P6

INTERVENTIONS:
Drug: scopolamine patch — Group I (n=80): Will receive scopolamine patch placement on the skin behind the right ear 1 hour before initiation of the regional anesthesia for the duration of surgery. The time of the application of the patch will be recorded, and the time of the start of the surgery will be recorded. The last time point for evaluation of patient's nausea/vomiting will be when the patient arrives to the post anesthesia care unit. A member of the research team will remove the patch from the patient and properly dispose the patch upon arrival to the post anesthesia care unit.
  Other Names: Transderm-Scop; Scopace; Maldemar
  Arms: scopolamine patch; scopolamine patch + acupressure point P6
Device: acupressure point P6 — Group II (n=80): Will receive acupressure point P6 stimulation. This is a stimulation of the chi channel at the master of the heart (MH8 position) at the small depression of the volar surface of the distal right forearm just above the crest of the wrist. The device will be put on the patients in the operating room prior to administration of the regional anesthesia and will be removed after the cesarean section is complete. The device will be removed from the patient in the operating room, before the patient is transported to the recovery room. Patients will receive continuous stimulation at a level that is comfortable for her prior to administration of the standardized regional anesthesia.
  Arms: acupressure point P6; scopolamine patch + acupressure point P6

SUMMARY:
The purpose of this study is to compare the effectiveness of reducing intra-cesarean section nausea and vomiting with regional anesthesia in subjects who will receive scopolamine patch with acupressure point P6 stimulation versus subjects that receive just scopolamine patch versus subjects that receive just acupressure point P6 stimulation.

DETAILED DESCRIPTION:
Nausea and vomiting are very common and unpleasant events experienced during cesarean section under regional anesthesia and in the postoperative period following cesarean section. These side effects are distressing for both the parturient and her family. In addition, intraoperative vomiting causes significant challenges for the surgeon, such as increased procedure length, increased risk of bleeding, increased risk of gastric content aspiration, and potential surgical trauma.

To combat the nausea and vomiting seen in all above anesthetic modalities, but to a greater degree in regional anesthesia, a number of pharmacological interventions are currently used with varying degrees of effectiveness in the perioperative period. These medications come from a wide range of drug classes including serotonin and dopamine receptor antagonists, corticosteroids, antihistamines, sedatives and anticholinergics.

In our study, we would like to compare the effectiveness of antiemetic agents or technique which cause less severe adverse reactions to the mother and her fetus. Out of the available pharmacological agents for reduction of intra-cesarean section nausea and vomiting, transdermal scopolamine patch is one of the safest medications. We would like to compare the effectiveness of the transdermal scopolamine patch with acupressure point P6 stimulation versus just transdermal scopolamine patch versus just acupressure point P6 stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ages 18 to 45
2. Subjects with ASA Class I or II
3. Subjects with elective primary or repeat cesarean delivery
4. Subjects who receive spinal and/or epidural anesthesia
5. English and non-English speaking subjects will be included in the study

Exclusion Criteria:

1. Female subjects <18 years of age
2. Subjects requiring emergent cesarean delivery
3. Gestational age < 37 weeks
4. History of placenta accreta
5. Multiple gestation pregnancy
6. ASA status III or higher
7. Current history of pregnancy induced hypertension, pre-eclampsia, or eclampsia
8. History of any chronic medication use (other than prenatal vitamins), including inhaler medications
9. Current urinary tract infection, pneumonia, or otitis media
10. Coagulopathies or skin infections overlying the spine
11. History of open angle glaucoma, seizures or psychosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Cohen, MD, Principal Investigator — Robert Wood Johnson University Hospital
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkins JL, Koonin LM, Palmer SK, Gibbs CP. Anesthesia-related deaths during obstetric delivery in the United States, 1979-1990. Anesthesiology. 1997 Feb;86(2):277-84. doi: 10.1097/00000542-199702000-00002. PMID 9054245
- [Background] Ezri T, Szmuk P, Evron S, Geva D, Hagay Z, Katz J. Difficult airway in obstetric anesthesia: a review. Obstet Gynecol Surv. 2001 Oct;56(10):631-41. doi: 10.1097/00006254-200110000-00022. PMID 11590314
- [Background] Malvasi A, Tinelli A, Stark M, Pontrelli G, Brizzi A, Wetzl RG, Benhamou D. Low-dose sequential combined spinal-epidural anaesthesia in elective Stark caesarean section: a preliminary cohort study. Eur Rev Med Pharmacol Sci. 2010 Mar;14(3):215-21. PMID 20391961
- [Background] Afolabi BB, Lesi FE. Regional versus general anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004350. doi: 10.1002/14651858.CD004350.pub3. PMID 23076903
- [Background] Riley ET, Cohen SE, Macario A, Desai JB, Ratner EF. Spinal versus epidural anesthesia for cesarean section: a comparison of time efficiency, costs, charges, and complications. Anesth Analg. 1995 Apr;80(4):709-12. doi: 10.1097/00000539-199504000-00010. PMID 7893022
- [Background] Balki M, Carvalho JC. Intraoperative nausea and vomiting during cesarean section under regional anesthesia. Int J Obstet Anesth. 2005 Jul;14(3):230-41. doi: 10.1016/j.ijoa.2004.12.004. PMID 15935649
- [Background] Paranjothy S, Griffiths JD, Broughton HK, Gyte GM, Brown HC, Thomas J. Interventions at caesarean section for reducing the risk of aspiration pneumonitis. Cochrane Database Syst Rev. 2014 Feb 5;2014(2):CD004943. doi: 10.1002/14651858.CD004943.pub4. PMID 24497372
- [Background] Flake ZA, Linn BS, Hornecker JR. Practical selection of antiemetics in the ambulatory setting. Am Fam Physician. 2015 Mar 1;91(5):293-6. PMID 25822385
- [Background] Golembiewski J, Chernin E, Chopra T. Prevention and treatment of postoperative nausea and vomiting. Am J Health Syst Pharm. 2005 Jun 15;62(12):1247-60; quiz 1261-2. doi: 10.1093/ajhp/62.12.1247. PMID 15947124
- [Background] Apfel CC, Zhang K, George E, Shi S, Jalota L, Hornuss C, Fero KE, Heidrich F, Pergolizzi JV, Cakmakkaya OS, Kranke P. Transdermal scopolamine for the prevention of postoperative nausea and vomiting: a systematic review and meta-analysis. Clin Ther. 2010 Nov;32(12):1987-2002. doi: 10.1016/j.clinthera.2010.11.014. PMID 21118734
- [Background] Renner UD, Oertel R, Kirch W. Pharmacokinetics and pharmacodynamics in clinical use of scopolamine. Ther Drug Monit. 2005 Oct;27(5):655-65. doi: 10.1097/01.ftd.0000168293.48226.57. PMID 16175141
- [Background] Lee A, Fan LT. Stimulation of the wrist acupuncture point P6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003281. doi: 10.1002/14651858.CD003281.pub3. PMID 19370583
- [Background] Allen TK, Habib AS. P6 stimulation for the prevention of nausea and vomiting associated with cesarean delivery under neuraxial anesthesia: a systematic review of randomized controlled trials. Anesth Analg. 2008 Oct;107(4):1308-12. doi: 10.1213/ane.0b013e31816d1864. PMID 18806045
- [Background] Quinla JD, Hill DA. Nausea and vomiting of pregnancy. Am Fam Physician. 2003 Jul 1;68(1):121-8. PMID 12887118
- [Background] Belluomini J, Litt RC, Lee KA, Katz M. Acupressure for nausea and vomiting of pregnancy: a randomized, blinded study. Obstet Gynecol. 1994 Aug;84(2):245-8. PMID 8041539
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Started | 80 | 80 | 80
Completed | 80 | 80 | 80
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6 | Total
Number analyzed (Participants) | 80 | 80 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is missing for one of the participants.
  years
    number analyzed (Participants) | 80 | 79 | 80 | 239
    (all) | 32.78 (4.98) | 31.32 (5.30) | 32.16 (4.87) | 31.94 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 80 | 240
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: inches] — Population: Height measurement is missing for one observation.
  inches
    number analyzed (Participants) | 80 | 80 | 79 | 239
    (all) | 64.7 (5) | 64.3 (4.5) | 64.2 (3.6) | 64.4 (4.4)
Weight [Mean (Standard Deviation); unit: lbs] | 188.11 (34.10) | 179.17 (30.20) | 184.51 (40.17) | 183.93 (35.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Nausea
Description: The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea at any point during the surgical procedure in each group.
Time Frame: Throughout the entire surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
Participants | 40 | 39 | 46
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: Percent experiencing nausea equal between groups; Test type: Other; p = 0.98, Chi-squared — Bonferroni-adjusted P-value, calculated as two times the nominal p-value because there are two primary outcomes; d.f.=2

2. Primary Outcome: Number of Patients With Vomiting
Description: The investigators will perform objective assessments of whether or not the patients have vomited during the procedure. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: Throughout the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
Participants | 24 | 25 | 31
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: Percent experiencing vomiting equal across groups; Test type: Other; p = 0.90, Chi-squared — Bonferroni-adjusted P-value, calculated as two times the nominal p-value because there are two primary outcomes; d.f.=2

3. Secondary Outcome: Satisfaction With Intraoperative Antiemetic Treatment
Description: Patients are asked their nausea and vomiting treatment satisfaction (0 = Not Satisfied, 10 = Extremely Satisfied). Patients are also asked their overall satisfaction with the procedure (0 = Not Satisfied, 10 = Extremely Satisfied).
Time Frame: Throughout the surgical procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
units on a scale | 9.29 (1.39) | 8.96 (9.59) | 9.59 (9.83)
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Test type: Other — Null hypothesis: Mean scores equal across treatment groups; p = 0.026, ANOVA

4. Secondary Outcome: Level of Nausea After the Administration of the Regional Anesthesia Medications
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) after the administration of the regional anesthesia medications. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: From administration of anaesthesia until eversion of uterus
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
units on a scale | 2.71 (4.02) | 2.57 (3.84) | 2.84 (3.99)
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Test type: Other — Null hypothesis: means equal across treatment groups; p = 0.91, ANOVA

5. Secondary Outcome: Level of Nausea After Eversion of the Uterus
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) after eversion of the uterus. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: After eversion of the uterus until replacement of the uterus
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
units on a scale | 1.28 (3.00) | 1.09 (2.82) | 1.40 (3.27)
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: means equal across treatment groups; Test type: Other; p = 0.80, ANOVA

6. Secondary Outcome: Level of Nausea After Replacement of the Uterus
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) after replacement of the uterus. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: After replacement of the uterus and to the next 15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
units on a scale | 2.19 (3.50) | 2.19 (3.78) | 2.51 (3.91)
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: means equal across treatment groups; Test type: Other; p = 0.82, ANOVA

7. Secondary Outcome: Level of Nausea Upon Arrival to the Post-operative Recovery Room
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) upon arrival to the post-operative recovery room. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: 15 minutes after replacement of the uterus to arrival at post-anaesthesia care unit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
units on a scale | 0.18 (1.11) | 0.25 (1.36) | 0.23 (1.42)
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: means equal across treatment groups; Test type: Other; p = 0.93, ANOVA

8. Secondary Outcome: Number of Patients With Vomiting After the Administration of the Regional Anesthesia Medications
Description: Objective assessments of whether or not the patients have vomited at this point in the surgical procedure will be done. The investigators will analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: After the administration of the regional anesthesia medications until eversion of the uterus
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
Participants | 20 | 15 | 20
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Test type: Other — Null hypothesis: percent of vomiting equal across treatment groups; p = 0.55, Chi-squared; d.f.=2

9. Secondary Outcome: Number of Patients With Vomiting After Eversion of the Uterus
Description: as for outcome 8
Time Frame: After eversion of to replacement of the uterus
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 80
Participants | 8 | 6 | 9
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: percent of vomiting equal across treatment groups; Test type: Other; p = 0.71, Chi-squared; d.f.=2

10. Secondary Outcome: Number of Patients With Vomiting After Replacement of the Uterus
Description: as for outcome 8
Time Frame: After replacement of the uterus and for next 15 minutes
Population: Missing information on one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 80 | 80 | 79
Participants | 10 | 15 | 12
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: percent of vomiting equal across treatment groups; Test type: Other; p = 0.55, Chi-squared; d.f.=2

11. Secondary Outcome: Number of Patients With Vomiting Upon Arrival to the Post-operative Recovery Room
Description: as for outcome 8
Time Frame: From 15 minutes after replacement of the uterus until arrival at the post-anaesthesia care unit
Population: Missing information on four participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
Number analyzed (Participants) | 79 | 80 | 77
Participants | 1 | 1 | 4
Statistical Analysis 1: Comparison: Scopolamine Patch vs Acupressure Point P6 vs Scopolamine Patch + Acupressure Point P6; Null hypothesis: percent of vomiting equal across treatment groups; Test type: Other; p = 0.20, Chi-squared; d.f.=2

ADVERSE EVENTS:
Time Frame: Intraoperative
Arm/Group | Scopolamine Patch | Acupressure Point P6 | Scopolamine Patch + Acupressure Point P6
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02960113/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02960113/SAP_001.pdf
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02960113/ICF_002.pdf